CLINICAL TRIAL: NCT02074618
Title: Impact of Physical Therapy on Functional Capacity and Quality of Patients With Chronic Kidney Disease
Brief Title: Physiotherapy in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional Publico do Araguaia (Other)
Responsible Party: Principal Investigator, Georgia Miranda Tomich, 1- Physiotherapist, Master in Rehabilitation Sciences, Coordinator of the Center for Study and Research of the Hospital Regional Publico do Araguaia, Redenção, PA, Brazil, Hospital Regional Publico do Araguaia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMT2013
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Disease.
Keywords: Physical Therapy.; Exercise.; Rehabilitation.; Renal Insufficiency.; Quality of life.
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Renal Insufficiency | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Exercise (Experimental): The program of physical exercise was a resistance and aerobic training, initiated at low intensity and with a slow progressing according to the patient's tolerance. In aerobic exercise, for greater effectiveness of the training, the literature recommends moderate intensity, which corresponds with 50 to 70% of the maximum heart rate. Patients were instructed to keep the most constant as possible the speed during exercise on treadmill or cycle ergometer. For muscle strengthening exercises, the number of repetitions varied from 1 to 4 sets of 10 to 15 repetitions.
  Interventions: Other: Physical exercise.

INTERVENTIONS:
Other: Physical exercise. — Physical exercises were held three times a week on alternate days to hemodialysis sessions, with duration of 45 to 90 minute, supervised by a physiotherapist. In all the sessions the following measurements were performed: body weight and blood pressure, heart rate and peripheral oxygen saturation in the pre, during and post session. The exercises were: heating and stretching during 5 minutes, followed by aerobic physical exercise on treadmill and/or bike (about 30 minutes), muscle strengthening exercises (15 to 20 minutes), cooling and stretching (5 minutes). The time for aerobic and strengthening varied according to the tolerance of the patient. The resistance exercises have been conducted for the major muscle groups of the lower limbs.

SUMMARY:
The purpose of this study was to evaluate the effects of physiotherapy based on the practice of supervised exercise on functional capacity and life quality of patients with chronic kidney disease.

DETAILED DESCRIPTION:
This quasi-experimental study, with repeated measures design, was held in the ambulatory of physical therapy, in a public hospital, which serves 15 cities in the South and Southeast of the state of Pará (Brazil) and has structure of hemodialysis, outpatient, wards and intensive care units.

For inclusion in the study, the patient should have age over 18 years, make part of the hospital's hemodialysis program, receive medical prescription for practice of physical activity, and sign an informed consent. The present study was carried out in accordance with National Health Council Resolution nº 196/96 of the Brazilian Ministry of Health, and approved by the Research Ethics Committee of the Tropical Medicine Foundation of Tocantins (protocol No. 023/2011).

Contraindications to physical activity practice were considered exclusion criteria: recent myocardial infarction; uncontrolled arrhythmias; uncontrolled hypertension (systolic blood pressure > 200mmHg and diastolic blood pressure > 120mmHg); unstable angina; severe decompensate diabetes (blood glucose > 300 mg/dL); left ventricle dysfunction; presence of neurological or motor dysfunction that was impeditive for implementation of the protocol of physical activity. Other exclusion criteria were: tumor; pregnancy; stopping treatment in the first 6 weeks for more than 3 consecutive sessions.

At the beginning of each exercise session, if the patient had any symptoms that prevented the exercises performance, it was canceled. After the start of the session, break criteria were considered: the account of intense physical tiredness, chest pain, dizziness, paleness, syncope, pre-syncope, dyspnea disproportionate to the intensity of the effort, arrhythmia and hypotension or hypertensive response. When any of these symptoms was detected, the patient was transferred to hemodialysis service for medical evaluation.

The data were analyzed in the program Statistical Package for the Social Sciences (SPSS) version 20.0 for Windows and are expressed as mean ± standard deviation. The Wilcoxon test was used for comparison of the averages of the values obtained at the beginning of the program and in reevaluation after six weeks. In all analyses, a statistical significance level of 0.05 was considered.

Initially, an interview was conducted with the patient, to collect data as the previous and current history, co-morbidities, medications, postural changes, vital signs. In the initial contact and after six weeks, in addition to anthropometric data, the following evaluations were carried out in order to assess the effects of the exercise protocol:

* Six-minute walk test (6MWT): measurement of functional capacity, which was carried out following the recommendations from the American Thoracic Society. This test has already been used in patients with chronic kidney disease in different studies found in literature; Reboredo et al. found a strong correlation between the distance obtained in 6MWT and peak oxygen consumption, suggesting that this test is a simple and inexpensive alternative for assessing the functional capacity of patients with chronic kidney disease who are undergoing hemodialysis treatment.
* Sit-to-stand test: test initially described as a measure of strength of lower extremity, it is currently also considered a balancing test and has already been validated in patients with chronic kidney disease.
* Quality of life assessment: the generic questionnaire Short-form 36 (SF36), translated into Portuguese was used for evaluation of life quality. Johansen et al. considered that the physical component of the SF36 is valid to assess physical performance in patients with chronic kidney disease on hemodialysis. Other authors such as Bohlke et al. and Arenas et al. used this test in patients with chronic kidney disease.

In all the sessions the following measurements were performed: body weight and blood pressure, heart rate and peripheral oxygen saturation in the pre, during and post session. The exercises were: heating and stretching during 5 minutes, followed by aerobic physical exercise on treadmill and/or bike (about 30 minutes), muscle strengthening exercises (15 to 20 minutes), cooling and stretching (5 minutes). The time for aerobic and strengthening varied according to the tolerance of the patient. The resistance exercises have been conducted for the major muscle groups of the lower limbs. All these activities were performed under the supervision and guidance of a physiotherapist responsible for research. The session had total duration of about 60 minutes - 5 minutes for the daily assessment of the patient, and the 55 minutes remaining divided among the exercises.

The program of resistance and aerobic training was initiated at low intensity and with a slow progressing according to the patient's tolerance. In aerobic exercise, for greater effectiveness of the training, the literature recommends moderate intensity, which corresponds with 50 to 70% of the maximum heart rate and the score of Borg scale around. These were the criteria considered in this study. Patients were instructed to keep the most constant as possible the speed during exercise on treadmill or cycle ergometer. For muscle strengthening exercises, the number of repetitions varied from 1 to 4 sets of 10 to 15 repetitions.

The exercises were held three times a week on alternate days to hemodialysis sessions. According to the literature, it is recommend at least three weekly sessions of 45 to 90 minute supervised exercises.

The equipment for carrying out the exercises and evaluations were blood pressure device, stethoscope, pulse oximeter, treadmill, cycle ergometry, mats, pillows, lingbar, dumbbells, elastic bands (Theraband ®), shin pads, therapeutic balls, chairs, two steps stairs.

Data collection was performed by only one physiotherapist. After the end of the period of data collection, the patients remained in rehabilitation service to continue the practice of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* To be age over 18 years.
* To make part of the hospital's hemodialysis program.
* To receive medical prescription for practice of physical activity and sign an informed consent.

Exclusion Criteria:

* Recent myocardial infarction.
* Uncontrolled arrhythmias.
* Uncontrolled hypertension (systolic blood pressure > 200mmHg and diastolic blood pressure > 120mmHg).
* Unstable angina.
* Severe decompensate diabetes (blood glucose > 300 mg/dL).
* Left ventricle dysfunction.
* Presence of neurological or motor dysfunction that was impeditive for implementation of the protocol of physical activity.
* Tumor.
* Pregnancy.
* Stopping treatment in the first 6 weeks for more than 3 consecutive sessions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Effect of physiotherapy on distance obtained with six-minute walk test as a measurement of functional capacity in patients with chronic kidney disease. | Six weeks.
  Six-minute walk test is a measurement of functional capacity, which was carried out following the recommendations from the American Thoracic Society. This test has already been used in patients with chronic kidney disease in different studies found in literature.
Effect of physiotherapy on number of repetitions obtained with sit-to-stand test as a measurement of functional capacity in patients with chronic kidney disease. | Six weeks.
  Sit-to-stand test is test initially described as a measure of strength of lower extremity, it is currently also considered a balancing test and has already been validated in patients with chronic kidney disease.

SECONDARY OUTCOMES:
Effect of physiotherapy on life quality of patients with chronic kidney disease. | Six weeks.
  Short-form 36 (SF36) is a generic questionnaire, translated into Portuguese was used for evaluation of life quality and already used in patients with chronic kidney disease on hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia M Tomich, Master, Principal Investigator — Hospital Regional Publico do Araguaia